CLINICAL TRIAL: NCT02397278
Title: Intra Articular Injections With Platelet Rich Plasma in Patients With Juvenile Osteochondritis Dissecans of the Knee: Does it Help? A Clinical and Magnetic Resonance Imaging (MRI) Study.
Brief Title: Intra Articular Injections With Platelet Rich Plasma in Patients With Juvenile Osteochondritis Dissecans of the Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Terumo BCT (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-2797
Record Dates: First submitted 2015-02-24; First posted 2015-03-24 (Estimated); Results first posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Osteochondritis Dissecans
MeSH Terms: conditions — Osteochondritis Dissecans

STUDY DESIGN:
Intervention Model Description: Arm 1- Conservative Treatment Arm 2- PRP Injections
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Platelet rich plasma (PRP) (Active Comparator): Patients will receive three PRP injections into the symptomatic knee; they will also be fitted with a hinged brace locked in extension, with weight bearing as tolerated and crutches for those with pain upon weight bear, complete rest from impact activities with progression to weight bearing as tolerated for 6 weeks, and then followed according to the Sports Medicine department's protocol for OCD.
  Interventions: Drug: Platelet rich plasma (PRP)
- Conventional therapy (No Intervention): Patients will be fitted with a hinged brace locked in extension, with weight bearing as tolerated and crutches for those with pain upon weight bear, complete rest from impact activities with progression to weight bearing as tolerated for 6 weeks, and then followed according to the Sports Medicine department's protocol for OCD.

INTERVENTIONS:
Drug: Platelet rich plasma (PRP) — Patient will receive 3 intra articular injections with autologous PRP in the affected knee and then follow conventional therapy.
  Other Names: autologous PRP
  Arms: Platelet rich plasma (PRP)

SUMMARY:
This study plans to learn more about ways to treat a joint problem in the knee called Juvenile Osteochondritis Dissecans (OCD). The goal of this study is to see if injecting platelet-rich plasma (PRP) into the knee can help knee cartilage heal faster, and will try to determine whether the injections lead to improvements in pain, performance of activities of daily living, improvements is sports activities and overall function and symptoms reduction. The investigators will compare PRP treatment to conservative therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age 10 - 17 inclusive with open physis confirmed by MRI
2. Documented symptomatic stable juvenile osteochondritis dissecans of the knee based on MRI without changes of osteoarthritis and no prior history of knee surgery.
3. The patient must be able to hold still without sedation for approximately 1 hour and must pass MRI screening evaluation for retained metal.
4. Patients with Di Paola stage 1 or 2 lesions

Exclusion Criteria:

1. Patients with polyarticular disease.
2. Patients with blood disorders (Blood disorders (thrombopathy, thrombocytopenia, anemia with hemoglobin <9g/dL). Only those patients with a positive history of blood disorders will have a Complete Blood Count (CBC) performed a week prior to inclusion in the study.
3. Patients who had intra-articular treatment with steroids within 3 months
4. Patients who are pregnant or nursing at the time of consent.
5. Patients with inflammatory arthritic conditions (e.g. rheumatoid arthritis)
6. Non-English speaking patients. (Scores used for evaluation have not been validated in Spanish)
7. Patients who had previous knee surgery
8. Additional disabilities in any of the lower limbs that would interfere with any of the clinical assessments.
9. Chronic use of NSAID (defined as taking non-steroidal anti-inflammatory drug) regularly every week for the last 6 months), steroids or chemotherapy drugs
10. Treatment with NSAIDs within 15 days prior to randomization in this study
11. Patients with a BMI over 30. Due to the fact that this study utilizes an injection technique which may be inaccurate in obese subjects.
12. Patients with a prolongation of bleeding time, e.g. those receiving anticoagulant drug therapy
13. Patients with a contraindication to MRI including: patients with cardiac pacemaker or non-approved intracranial vascular clip, and those with orthopedic hardware as the resulting artifact can complicate interpretation
14. Patients with acute or chronic renal failure
15. Patients with a previous anaphylactic reaction to gadolinium enhanced MRI.
16. Patients with Di Paola stage 3 or 4 lesions

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2020-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fadell, MD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Platelet Rich Plasma (PRP) | Conventional Therapy
Started | 7 | 8
Completed | 6 | 5
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Deemed ineligible following surgery | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Platelet Rich Plasma (PRP) | Conventional Therapy | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 8 | 15
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 12 [10 to 13] | 11.335 [10 to 14] | 11.6 [10 to 14]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 4 | 7 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 7 | 6 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 8 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Greater Cartilage Healing Measured by Glycosaminoglycan Content on dGEMRIC MRI
Description: Measured by dGEMRIC MRI
Time Frame: 6 months
Population: This outcome measure for post-contrast dGEMRIC studies was not collected. The protocol was amended to include non-contrast studies due to difficulty recruiting patients.
Arm/Group | Platelet Rich Plasma (PRP) | Conventional Therapy
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Improvement in Pain, Performance and Overall Function: IKDC
Description: Measured by the Pediatric IKDC survey results. The International Knee Documentation Committee questionnaire measures knee function, Scores range from 1-100, with higher scores indicating a better outcome.
Time Frame: Baseline, 6 months, 12 months
Population: Not all participants were available for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Platelet Rich Plasma (PRP) | Conventional Therapy
Number analyzed (Participants) | 8 | 5
score on a scale
  Baseline | 48 (21) | 52 (34)
  Month 6 | 86 (21) | 84 (20)
  Month 12 | 84 (18) | 90 (9)

3. Other Pre Specified Outcome: dGemric MRI Findings Correlate With Measures of Functional Recovery and Symptom Reduction.
Description: Measured by the results of the dGEMRIC MRI and the IKDC and KOOS survey results
Time Frame: 6 months
Reporting Status: Not Posted

4. Secondary Outcome: Improvement in Pain, Performance and Overall Function: KOOS, Baseline
Description: Measured by the KOOS survey results. The Knee injury and Osteoarthritis Outcome Score (KOOS) measures patient reported knee function and quality of life. Possible scores range from 0 to 100, with higher scores indicating a better outcome.
Time Frame: Baseline
Population: Not all participants were available for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Platelet Rich Plasma (PRP) | Conventional Therapy
Number analyzed (Participants) | 8 | 5
score on a scale
  Pain Subscale | 56.8 (21.6) | 50.0 (24.6)
  Symptoms Subscale | 67.3 (24.7) | 65.0 (17.0)
  Activities of Daily Living Subscale | 70.1 (24.5) | 60.7 (25.2)
  Sport Subscale | 23.8 (21.1) | 30.7 (42.2)
  Quality of Life Subscale | 43.1 (19.9) | 28.3 (20.3)

5. Secondary Outcome: Improvement in Pain, Performance and Overall Function: KOOS, 6 Months
Description: as for outcome 4
Time Frame: 6 Months
Population: Not all participants were available for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Platelet Rich Plasma (PRP) | Conventional Therapy
Number analyzed (Participants) | 6 | 4
score on a scale
  Pain Subscale | 90.6 (15.6) | 91.4 (10.6)
  Symptoms Subscale | 84.6 (5.4) | 89.3 (12.3)
  Activities of Daily Living Subscale | 95.8 (10.2) | 96.6 (3.9)
  Sport Subscale | 88.1 (29.2) | 69.6 (40.6)
  Quality of Life Subscale | 68.1 (22.6) | 53.1 (32.5)

6. Secondary Outcome: Improvement in Pain, Performance and Overall Function: KOOS, 12 Months
Description: as for outcome 4
Time Frame: 12 Months
Population: Not all participants were available for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Platelet Rich Plasma (PRP) | Conventional Therapy
Number analyzed (Participants) | 8 | 4
score on a scale
  Pain Subscale | 85.9 (16.4) | 93.8 (8.3)
  Symptoms Subscale | 92.9 (5.0) | 94.0 (10.3)
  Activities of Daily Living Subscale | 90.5 (13.1) | 99.2 (1.3)
  Sport Subscale | 75.6 (30.8) | 91.7 (14.4)
  Quality of Life Subscale | 56.9 (24.2) | 75.0 (14.4)

ADVERSE EVENTS:
Time Frame: 12 Months
Arm/Group | Platelet Rich Plasma (PRP) | Conventional Therapy
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 0/7 | 0/8

LIMITATIONS AND CAVEATS:
The 12 month time point for primary and secondary outcome measures was mistakenly omitted from the original registration. This has been corrected to align with the currently approved protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-28): https://cdn.clinicaltrials.gov/large-docs/78/NCT02397278/Prot_SAP_000.pdf